CLINICAL TRIAL: NCT06447155
Title: The Impact of Continuous Versus Bolus Feeding in Neonates With Hypoxic Ischemic Encephalopathy Undergoing Therapeutic Hypothermia
Brief Title: Continuous Versus Bolus Feeding in Neonates With Hypoxic Ischemic Encephalopathy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, DİDEM ARMAN, Associate Professor, Istanbul Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IstanbulTRH-DArman-003
Record Dates: First submitted 2024-06-03; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Hypoxic Ischemic Encephalopathy of Newborn; Feeding Patterns
Keywords: Newborn; Hypoxic ischemic encephalopathy; Enteral feeding; Bolus; Continuous
MeSH Terms: conditions — Feeding Behavior; Hypoxia-Ischemia, Brain

STUDY DESIGN:
Intervention Model Description: The babies were randomized into three groups; Group 1.The neonates who received bolus feeding,Group 2. The neonates who received continuous feeding Group 3. The control group who were not fed during TH. The control group was composed of historical newborns. Three groups were compared in terms of demographic characteristics and clinical outcomes.
Who Masked: Participant, Investigator
Masking Description: Care provider decides the type of feeding according to the randomization list which were prepared via a website (http://www.randomizer.org)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The babies fed with bolus feeding during TH (Active Comparator): The babies were randomized into three groups; Group 1.The neonates who received bolus feeding,Group 2. The neonates who received continuous feeding Group 3. The control group who were not fed during TH. The control group was composed of historical newborns. Three groups were compared in terms of demographic characteristics and clinical outcomes.
  Interventions: Dietary Supplement: Bolus feeding
- The babies fed with continuous feeding during TH (Active Comparator): The babies were randomized into three groups; Group 1.The neonates who received bolus feeding,Group 2. The neonates who received continuous feeding Group 3. The control group who were not fed during TH. The control group was composed of historical newborns.Three groups were compared in terms of demographic characteristics and clinical outcomes.
  Interventions: Dietary Supplement: Continuous feeding
- The babies who were not fed (Placebo Comparator): The babies were randomized into three groups; Group 1.The neonates who received bolus feeding,Group 2. The neonates who received continuous feeding Group 3. The control group who were not fed during TH. The control group was composed of historical newborns.Three groups were compared in terms of demographic characteristics and clinical outcomes.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Bolus feeding — The babies fed with bolus feeding during TH composed this group
  Arms: The babies fed with bolus feeding during TH
Dietary Supplement: Continuous feeding — The babies fed with continuous feeding during TH composed this group
  Arms: The babies fed with continuous feeding during TH
Dietary Supplement: Placebo — The babies who were not fed during TH composed this group
  Arms: The babies who were not fed

SUMMARY:
Therapeutic hypothermia (TH) is accepted worldwide as a standard of care for infants born at or beyond 36 weeks gestational age with moderate-to-severe hypoxic ischaemic encephalopathy (HIE).

While central nervous system is the most affected organ system , multiorgan dysfunction including renal, pulmonary, cardiac, and/or gastrointestinal (GI) compromise is not infrequent. Although the process of 'cooling' itself is well defined, based on high-quality randomized controlled trials, there are few data to inform the provision of nutrition to infants with HIE during and soon after TH.However, breastfeeding plays a beneficial role in maintaining the structural and functional integrity of the gut. It may help to reduce systemic inflammatory response and positively regulates the microbiota. In many studies it is stated that enteral feeding during TH appears to be safe and feasible. There is insufficient evidence to choose the type of enteral feeding either bolus or continuous during TH.

The present study aimed to compare the impact of different types of enteral feeding in infants with HIE receiving TH.

DETAILED DESCRIPTION:
Objectives: The investigators aimed to evaluate the clinical consequences of different types of enteral nutrition during TH in babies with HIE.

Methods: This single-center, prospective randomized controlled trial (RCT) was conducted between June 2024 to June 2026 in Istanbul Research and Training Hospital. A cohort of 60 infants with HIE, born at 35 0/7 to 42 6/7 weeks of gestation who received TH were enrolled.

The infants enterally fed with bolus feeding during hypothermia (n =20), those who were fed continuously (n=20) constituted the study groups. The control group (n =20) was composed of neonates who were not fed. Infants were monitored for clinical consequences such as feeding intolerance, time to full enteral feeding, duration of hospitalization, necrotizing enterocolitis and mortality.

ELIGIBILITY:
Inclusion Criteria:

* The neonates with evidence of encephalopathy de¬fined by seizures or abnormalities on a modified Sarnat exam were enrolled. The hypoxic-ischemic injury was defined by 1. a pH of ≤ 7.0 and/or 2. base deficit >-16 mmol/L recorded in cord blood or blood gas obtained within the first hour postnatally or a pH of 7.0 - 7.15 and/or base deficit (-10-15.9) mmol/L with the presence of an acute perinatal event (cord prolapse, placental abruption, heart rate decelerations, severe fetal bradycardia). In cases where criteria 1 or 2 are met, with the presence of seizures or a diagnosis of moderate to severe encephalopathy according to the Sarnat & Sarnat classification based on neurological examination were treated with TH.

Exclusion Criteria: Infants with congenital malformation or hereditary metabolic diseases, infants whose enteral feeding was initiated before randomization and infants without lack of parental consent were excluded. The maternal and neonatal demographic characteristics and clinical outcomes were collected from medical records.

-

Ages: 0 Days to 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Development of Necrotizing enterocolitis (NEC) | From admission to NICU till postnatal 15th day or hospital discharge whichever came first
  The infants will be monitorized for NEC development

SECONDARY OUTCOMES:
Feeding intolerance | From admission to NICU till postnatal 15th day or hospital discharge whichever came first
  The infants will be monitorized for feeding intolerance
Time to full enteral feeding | From admission to NICU till postnatal 15th day or hospital discharge whichever came first
  The infants will be monitorized for feeding intolerance

CONTACTS AND LOCATIONS:
Locations (1):
- IstanbulTRH, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data sets generated during and/or analyzed during current study may be available from the corresponding author on reasonable request.

REFERENCES:
- [Background] Azzopardi DV, Strohm B, Edwards AD, Dyet L, Halliday HL, Juszczak E, Kapellou O, Levene M, Marlow N, Porter E, Thoresen M, Whitelaw A, Brocklehurst P; TOBY Study Group. Moderate hypothermia to treat perinatal asphyxial encephalopathy. N Engl J Med. 2009 Oct 1;361(14):1349-58. doi: 10.1056/NEJMoa0900854. PMID 19797281
- [Background] Jacobs SE, Berg M, Hunt R, Tarnow-Mordi WO, Inder TE, Davis PG. Cooling for newborns with hypoxic ischaemic encephalopathy. Cochrane Database Syst Rev. 2013 Jan 31;2013(1):CD003311. doi: 10.1002/14651858.CD003311.pub3. PMID 23440789
- [Background] Martin-Ancel A, Garcia-Alix A, Gaya F, Cabanas F, Burgueros M, Quero J. Multiple organ involvement in perinatal asphyxia. J Pediatr. 1995 Nov;127(5):786-93. doi: 10.1016/s0022-3476(95)70174-5. PMID 7472837
- [Background] Sharma S, Kallesh A, Aradhya AS, Diggikar S, Veeraiah PS, Subbareddy NN, Walikar S, Reddy IV, Sarji D, Venkatagiri P. Feasibility of Minimal Enteral Nutrition During Therapeutic Hypothermia for Perinatal Asphyxia: A Five-Year Multicenter Experience from South India. Indian J Pediatr. 2023 May;90(5):513-515. doi: 10.1007/s12098-022-04456-x. Epub 2023 Jan 16. PMID 36642779
- [Background] Kumar J, Anne RP, Meena J, Sundaram V, Dutta S, Kumar P. To feed or not to feed during therapeutic hypothermia in asphyxiated neonates: a systematic review and meta-analysis. Eur J Pediatr. 2023 Jun;182(6):2759-2773. doi: 10.1007/s00431-023-04950-0. Epub 2023 Apr 4. PMID 37014443